CLINICAL TRIAL: NCT02317510
Title: Combined Spinal Epidural Anesthesia and General Anesthesia for Laparoscopic Cholecystectomy: a Prospective, Randomized Study
Brief Title: Combined Spinal Epidural Anesthesia and General Anesthesia for Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lütfiye Nuri Burat Government Hospital (Other Government)
Collaborators: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, TURGUT DONMEZ, Medical Doctor, General Surgeon, Lütfiye Nuri Burat Government Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HASEKI-156
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Gall Stone Disease; Polyp
Keywords: Combined anesthesia; General anesthesia; Laparoscopic cholecystectomy
MeSH Terms: conditions — Polyps | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): Laparoscopic cholecystectomy in General Anesthesia
  Interventions: Procedure: combined anesthesia
- group 2 (Active Comparator): Laparoscopic cholecystectomy in combined anesthesia (Spino epidural).
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: combined anesthesia — Combined Spinal Epidural Anesthesia for laparoscopic cholecystectomy
  Arms: group 1
Procedure: general anesthesia — General anesthesia for laparoscopic cholecystectomy
  Arms: group 2

SUMMARY:
The aim of this study was to compare general anesthesia (GA) and combined (epidural and spinal) anesthesia (CA) for laparoscopic cholecystectomy. General anesthesia is a gold standard for laparoscopic cholecystectomy(LC). The use of combined anesthesia may offer several advantages over general anesthesia.

Fifty patients will be randomly assigned to either the CA LC (25 patients) or GA LC (25 patients). All patients has symptomatic gall stone disease or polyp of gall bladder. Intraoperative events related to combined anesthesia , postoperative complications, pain score and duration of operation time will record.

DETAILED DESCRIPTION:
Objective of study : The aim of this study was to compare general anesthesia (GA) and combined (epidural and spinal) anesthesia (CA) for laparoscopic cholecystectomy. General anesthesia is a gold standard for laparoscopic cholecystectomy(LC). The use of combined anesthesia may offer several advantages over general anesthesia.

Material and methods : Fifty patients will be randomly assigned to either the CA LC (25 patients) or GA LC (25 patients). All patients has symptomatic gall stone disease or polyp of gall bladder. Intraoperative events related to combined anesthesia : abdominal discomfortable, shoulder pain, abdominal pain, nausea, anxiety, dermatomal level of sensory blockade, respiratory depression. We compare between two group; shoulder pain, postoperative complications, pain score, duration of operation time and length of hospital stay.

Fifty patients will select prospectively for LC, under low pressure (10 mm Hg) pneumoperitoneum and under combined anesthesia and general anesthesia. Spinal anaesthesia was performed at L1-L2 interspace using 2 ml of 0.5% (10 mg) hyperbaric Bupivacaine mixed with 0.5ml (25 micrograms) of Fentanyl. Epidural catheter was inserted at L1- L2 interspace too.

ELIGIBILITY:
Inclusion Criteria:

* Gall stone disease, polyp

Exclusion Criteria:

* Gall bladder cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Donmez, operator MD, Principal Investigator — Lutfiye NBGH
Locations (1):
- Lutfiye NBGH, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Bessa SS, Katri KM, Abdel-Salam WN, El-Kayal el-SA, Tawfik TA. Spinal versus general anesthesia for day-case laparoscopic cholecystectomy: a prospective randomized study. J Laparoendosc Adv Surg Tech A. 2012 Jul-Aug;22(6):550-5. doi: 10.1089/lap.2012.0110. Epub 2012 Jun 11. PMID 22686181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical clinic
Groups:
- Group 2: Laparoscopic cholecystectomy in combined anesthesia (Spinal epidural).
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Median (Standard Deviation); unit: years] | 46 (13.38) | 45.5 (13.60) | 46 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  Turkey | 25 | 24 | 49
BMI [Median (Standard Deviation); unit: kg/m^2] — BMI:Body Mass Index
  kg/m^2 | 28.66 (4.49) | 30.68 (3.59) | 29.55 (4.14)
ASA (American Society of Anesthesiologists scores) [Median (Full Range); unit: units on a scale] — The ASA score is a subjective assessment of a patient's overall health that is based on five classes (I to V).
  I- Patient is a completely healthy fit patient. II- Patient has mild systemic disease. III-Patient has severe systemic disease that is not incapacitating. IV-Patient has incapacitating disease that is a constant threat to life. V-A moribund patient who is not expected to live 24 hour with or without surgery.
  units on a scale | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Duration of Operation
Description: group 1:surgical operation time is 20 minutes minimum and maximum 55 minutes. Mean operation time 36.56 minutes group 2:surgical operation time is 24 minutes minimum and maximum 53 minutes. Mean operation time 30.75 minutes
Time Frame: up to 2 hours
Population: All patients have gall bladder disease who are between 18-90 years old.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
minutes | 36.56 (10.627) | 30.75 (7.502)

2. Secondary Outcome: Duration of Anaesthesia
Description: Group 1 minimum 42 minutes and maximum 83 minutes.mean duration of anaesthesia 60.17 and Group 2 minimum 45 minutes and maximum 82 minutes mean duration of anaesthesia 60.23
Time Frame: up to 2 hours
Population: All patients have gall bladder disease who are between 18-90 years old.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
minutes | 60.17 (10.73) | 60.23 (7.87)

3. Secondary Outcome: Post-operative Abdominal Pain 2nd Hour
Description: VAS score ;Explain to the person that each number describe the intensity of his pain. Number 0 describe very happy and no pain and no hurt at all. Number 1 hurts just a little bit. And as te numbers gradually increase pain will increase. Number 10 describes the worst pain in his life. Ask the patient to choose the number that best describes how he is feeling and his pain.
Time Frame: pain at postoperative 2nd hour
Population: All patients have gall bladder disease who are between 18-90 years old.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
units on a scale | 7 (0.71) | 1 (0.51)

4. Secondary Outcome: Post-operative Abdominal Pain 4th Hour
Description: as for outcome 3
Time Frame: pain at postoperative 4th hour
Population: All patients have gall bladder disease who are between 18-90 years old.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
units on a scale | 6 (0.71) | 2 (0.57)

5. Secondary Outcome: Post-operative Abdominal Pain 6th Hour
Description: VAS score;Explain to the person that each number describe the intensity of his pain. Number 0 describe very happy and no pain and no hurt at all. Number 1 hurts just a little bit. And as te numbers gradually increase pain will increase. Number 10 describes the worst pain in his life. Ask the patient to choose the number that best describes how he is feeling and his pain.
Time Frame: pain at postoperative 6th hour
Population: All patients have gall bladder disease who are between 18-90 years old.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
units on a scale | 4 (0.45) | 4 (0.6)

6. Secondary Outcome: Post-operative Abdominal Pain 12th Hour
Description: as for outcome 5
Time Frame: pain at postoperative 12th hour
Population: All patients have gall bladder disease who are between 18-90 years old.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
units on a scale | 3 (0.72) | 1 (0.46)

7. Secondary Outcome: Post-operative Abdominal Pain 24th Hour
Description: as for outcome 5
Time Frame: pain at postoperative 24th hour
Population: All patients have gall bladder disease who are between 18-90 years old.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
units on a scale | 2 (0.52) | 1 (0.50)

8. Primary Outcome: Post-operative Shoulder Pain
Description: Group 1 and Group 2 Post-operative shoulder pain
Time Frame: from end of the operation to postoperative 3 days
Population: All patients have gall bladder disease who are between 18-90 years old
Measure: Number; unit: participants
Groups:
- Group 2: Laparoscopic cholecystectomy in combined spinal epidural anaesthesia
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
participants
  shoulder pain yes | 15 | 6
  shoulder pain no | 10 | 18

9. Secondary Outcome: Intra-operative Shoulder Pain
Description: Group 1 and Group 2 Intra-operative shoulder pain
Time Frame: during operation time, up to 2 hours
Population: All patients have gall bladder disease who are between 18-90 years old.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
participants
  shoulder pain yes | 0 | 3
  shoulder pain no | 25 | 21

10. Secondary Outcome: Urinary Retention
Description: Group 1 and Group 2 Urinary retention
Time Frame: from end of the operation to postoperative 1 day
Population: All patients have gall bladder disease who are between 18-90 years old
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
participants
  urinary retention yes | 0 | 3
  urinary retention no | 25 | 21

11. Secondary Outcome: Nausea/Vomiting
Description: Group 1 and group 2 nausea/vomiting
Time Frame: from end of the operation to postoperative 1 day
Population: All patients have gall bladder disease who are between 18-90 years old.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
participants
  nausea/vomiting yes | 5 | 1
  nausea/vomiting no | 20 | 23

12. Secondary Outcome: Headache
Description: Group 1 and Group 2 Headache
Time Frame: from end of the operation to postoperative 3 days
Population: All patients have gall bladder disease who are between 18-90 years old.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 24
participants
  headache yes | 0 | 2
  headache no | 25 | 22

ADVERSE EVENTS:
Time Frame: December 2014-may 2015
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 21/25 | 16/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=25) | Group 2 (N=24)
mean vascular injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) — main vascular injury did not occur in both groups
embolism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) — embolism did not occur in both groups
choledocal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) — choledocal injury did not occur in both groups
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=25) | Group 2 (N=24)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
post-operative shoulder pain (Nervous system disorders) | 15 (15) | 6 (6) — post-operative shoulder pain;in both groups
Urinary retansion (Renal and urinary disorders) | 0 (0) | 3 (3) — Urinary retention;from end of the operation to postoperative 1 day
Nausea/vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) — Nausea/vomiting;intraoperative ve postoperative
Headache (Nervous system disorders) | 0 (0) | 2 (2) — Headache;from end of the operation to postoperative 3 days
intra-operative shoulder pain (Nervous system disorders) | 0 (0) | 3 (3) — intra-operative shoulder pain:during operation time, up to 2 hours

LIMITATIONS AND CAVEATS:
one patients had dural injury. Because of this that patient had released.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No